CLINICAL TRIAL: NCT03427775
Title: Assessment of Patient Outcomes After Shoulder Surgery After Implementation of a Multimodal Perioperative Management Protocol
Brief Title: Multimodal Analgesia After Shoulder Arthroscopy
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Nabil Elkassabany, Assistant Professor, University of Pennsylvania
Other Study IDs: 818312
Record Dates: First submitted 2018-01-29; First posted 2018-02-09 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Analgesia; Arthroscopy; Shoulder Joint
Keywords: multimodal analgesia; quality of recovery; quality of pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-MP3: before implementation of the multimodal analgesia protocol
- post-MP3: after implementation of the multimodal analgesia protocol
  Interventions: Combination Product: multimodal perioperative pain protocol (MP3)

INTERVENTIONS:
Combination Product: multimodal perioperative pain protocol (MP3) — administration of gabapentionoid, acetaminophen, non steroidal anti-inflammatory drugs around the clock in addition to the peripheral nerve block offered before surgery
  Groups: post-MP3

SUMMARY:
This proposal aims to measure the quality of recovery and quality of pain management after shoulder surgery before and after implementation of a multimodal pain protocol.

DETAILED DESCRIPTION:
Pain management after shoulder surgery remains to be a major challenge. Reliance on a single agent (most commonly opioids) results in increased incidence of side effects. Multimodal pain management refers to the use of multiple drugs that target different components of pain pathway.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Age 18-80
* Speaks and understands the English language
* Have a phone number
* Scheduled for shoulder arthroscopy

Exclusion Criteria:

* Inability to read or speak English
* Individuals outside of age range
* Pregnant women
* Persons under the jurisdiction of the Department of Corrections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled for shoulder arthroscopy
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
QOR-9 | 24 hours
  quality of recovery score using the QOR-9 instrument: it is a 9 item questionnaire with each question scoring from 0,1,2 with a total highest possible score of 18

SECONDARY OUTCOMES:
quality of pain management | 24 and 48 hours
  quality of pain management was measured using the revised american pain society patient oriented outcome questionnaire (APS-POQ-R). The questionnaire measures quality of pain management in 5 domains: 1- pain intensity 2- pain interference with activity and sleep 3- emotional side effects of uncontrolled pain ( affective scale). 4- patient perception of their pain management 5-side effects of pain treatment some questions answers are on a scale from 0-10. Ten is the maximum score and zero is the minimum score. other questions are listed as percentage with increments of 10% at a time (0%,10%, 20%, 30%..etc). each item/question is reported individually
amount of opioids | 24, 48 and 72 hours after surgery
  amount of opioids used converted to mg equivalent of oxycodone
QOR-9 | at 48 hours and 72 hours
  quality of recovery score using the QOR-9 instrument: it is a 9 item questionnaire with each question scoring from 0,1,2 with a total highest possible score of 18

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elkassabany NM, Wang A, Ochroch J, Mattera M, Liu J, Kuntz A. Improved Quality of Recovery from Ambulatory Shoulder Surgery After Implementation of a Multimodal Perioperative Pain Management Protocol. Pain Med. 2019 May 1;20(5):1012-1019. doi: 10.1093/pm/pny152. PMID 30113685